CLINICAL TRIAL: NCT00216931
Title: Treatment of Elevated Arterial Pulmonary Pressure With Inhaled Iloprost
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled after three years
Sponsor: Lund University Hospital (Other)
Collaborators: Bayer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-001551-11
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Persistent Pulmonary Hypertension; Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Iloprost

INTERVENTIONS:
Drug: iloprost

SUMMARY:
The purpose of this study is to determine if iloprost is effective in the treatment of elevated arterial pulmonary pressure in children with ventilator treated respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Elevated arterial pulmonary pressure
* GA > 24 GW
* 24-48 hours of age
* Ventilator treatment

Exclusion Criteria:

* Congenital anomalies
* Severe hypotension

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2006-05; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index
Cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Vineta Fellman, Professor, Principal Investigator — Lund University Hospital, Department of Pediatrics
Locations (1):
- University Hospital in Lund , Department of Pediatrics, Lund, Lund, Sweden